CLINICAL TRIAL: NCT03225326
Title: Efficacy of Anterior and Middle Superior Alveolar (AMSA) Nerve Block Anesthesia Obtained by Articaine Computer-controlled and Conventional Delivery
Brief Title: Effects of Articaine Computer-controlled and Conventional Delivery for Anterior and Middle Superior Alveolar Nerve Block for Tooth Extraction
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Bozidar Brkovic, DDS, MSc, PhD, Professor, DDS PhD Professor, University of Belgrade
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UBelgrade 784/2
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Local Anesthesia
Keywords: articaine; local anesthesia; AMSA
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: US Export: No

ARMS (2):
- Computer controlled 4% articaine delivery by Anaeject (Experimental)
  Interventions: Drug: Computer controlled 4% articaine delivery by Anaeject
- Conventional 4% articaine delivery by carpule syringe (Active Comparator)
  Interventions: Drug: Conventional 4% articaine delivery by carpule syringe

INTERVENTIONS:
Drug: Computer controlled 4% articaine delivery by Anaeject — Single dose of 0.6ml 4% articaine with epinephrine (1:100.000) delivered by computer controlled local anesthetic delivery system (Anaeject)
  Arms: Computer controlled 4% articaine delivery by Anaeject
Drug: Conventional 4% articaine delivery by carpule syringe — Single dose of 0.6ml 4% articaine with epinephrine (1:100.000) delivered by conventional syringe (carpule syringe).
  Arms: Conventional 4% articaine delivery by carpule syringe

SUMMARY:
The purpose of this study was to investigate and compare pulpal anesthesia and cardiovascular parameters obtained with 0.6 ml of 4% articaine with epinephrine (1:100.000) for anterior and middle superior alveolar nerve (AMSA) block performed by standard and computer-controlled delivery for maxillary teeth extraction.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1
* maxillary incisors canines or premolars indicated for extraction due to periapical pathology, root fracture or orthodontic treatment

Exclusion Criteria:

* allergies to local anesthetic solution ingredients, food and drugs
* alcohol and drugs abuse
* heavy tobacco smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Success of Pulpal Anesthesia for Central Incisive | after 1 hour
  Measured by pulp sensitivity to electrical pulp tester
Success of Pulpal Anesthesia for Lateral Incisive | after 1 hour
  Measured by pulp sensitivity to electrical pulp tester
Success of Pulpal Anesthesia for Canine | after 1 hour
  Measured by pulp sensitivity to electrical pulp tester
Success of Pulpal Anesthesia for First Premolar | after 1 hour
  Measured by pulp sensitivity to electrical pulp tester
Success of Pulpal Anesthesia for Second Premolar | after 1 hour
  Measured by pulp sensitivity to electrical pulp tester

SECONDARY OUTCOMES:
Onset Central Incisive | up to 8 minutes
  Measured by pulp sensitivity to electrical pulp tester
Onset Lateral Incisive | up to 8 minutes
  Measured by pulp sensitivity to electrical pulp tester
Onset Canine | up to 8 minutes
  Measured by pulp sensitivity to electrical pulp tester
Onset First Premolar | up to 8 minutes
  Measured by pulp sensitivity to electrical pulp tester
Onset Second Premolar | up to 8 minutes
  Measured by pulp sensitivity to electrical pulp tester
Duration Central Incisive | up to 60 minutes
  Measured by pulp sensitivity to electrical pulp tester
Duration Lateral Incisive | up to 60 minutes
  Measured by pulp sensitivity to electrical pulp tester
Duration Canine | up to 60 minutes
  Measured by pulp sensitivity to electrical pulp tester
Duration First Premolar | up to 60 minutes
  Measured by pulp sensitivity to electrical pulp tester
Duration Second Premolar | up to 60 minutes
  Measured by pulp sensitivity to electrical pulp tester
Systolic blood pressure | baseline
  Measured noninvasively in mm Hg
Systolic blood pressure at 5th minute | 5th minute
  Measured noninvasively in mm Hg
Systolic blood pressure at 10th minute | 10th minute
  Measured noninvasively in mm Hg
Systolic blood pressure at 15th minute | 15th minute
  Measured noninvasively in mm Hg
Systolic blood pressure at 30th minute | 30th minute
  Measured noninvasively in mm Hg
Diastolic blood pressure | baseline
  Measured noninvasively in mm Hg
Diastolic blood pressure at 5th minute | 5th minute
  Measured noninvasively in mm Hg
Diastolic blood pressure at 10th minute | 10th minute
  Measured noninvasively in mm Hg
Diastolic blood pressure at 15th minute | 15th minute
  Measured noninvasively in mm Hg
Diastolic blood pressure at 30th minute | 30th minute
  Measured noninvasively in mm Hg
Heart rate | baseline
  Measured noninvasively in beats per minute
Heart rate at 5th minute | 5th minute
  Measured noninvasively in beats per minute
Heart rate at 10th minute | 10th minute
  Measured noninvasively in beats per minute
Heart rate at 15th minute | 15th minute
  Measured noninvasively in beats per minute
Heart rate at 30th minute | 30th minute
  Measured noninvasively in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Marija Milić, Research Associate, Principal Investigator — School of Dental Medicine, University of Belgrade; Vladimir Biočanin, Assistant Professor, Principal Investigator — Faculty of Pharmacy and Health, University of Travnik, Bosnia and Herzegovina
Locations (1):
- School of Dental Medicine, University of Belgrade, Belgrade, Serbia